CLINICAL TRIAL: NCT00259636
Title: Zonisamide for Fibromyalgia & Migraine
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Logistical problems prevented enrollment
Sponsor: University of Pittsburgh (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Dawn Marcus, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EISAI 51-345-749
Record Dates: First submitted 2005-11-26; First posted 2005-11-29 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2011-05

CONDITIONS: Fibromyalgia; Migraine
MeSH Terms: conditions — Fibromyalgia; Migraine Disorders | interventions — Zonisamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: zonisamide — zonisamide 100 mg -300 mg daily vs placebo

SUMMARY:
Patients with fibromyalgia & migraine are randomized to receive zonisamide or placebo.

DETAILED DESCRIPTION:
Study was not conducted due to logistical problems

ELIGIBILITY:
Inclusion Criteria:

* 18-65 with fibromyalgia & migraine

Exclusion Criteria:

* allergy sulfa, liver or kidney disease, pregnant or not using contraception

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-08; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Visual analogue score | assessment measures at study enrollment (pre-treatment), and after 2, 4, and 8 weeks of treatment
  assessment measures at study enrollment (pre-treatment), and after 2, 4, and 8 weeks of treatment
Tender point count | assessment measures at study enrollment (pre-treatment), and after 2, 4, and 8 weeks of treatment
  assessment measures at study enrollment (pre-treatment), and after 2, 4, and 8 weeks of treatment
Headache index | assessment measures at study enrollment (pre-treatment), and after 2, 4, and 8 weeks of treatment
  assessment measures at study enrollment (pre-treatment), and after 2, 4, and 8 weeks of treatment

SECONDARY OUTCOMES:
Sleep efficiency | assessment measures at study enrollment (pre-treatment), and after 2, 4, and 8 weeks of treatment
  assessment measures at study enrollment (pre-treatment), and after 2, 4, and 8 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Marcus, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States